CLINICAL TRIAL: NCT03988725
Title: Nonalcoholic Steatohepatitis in HIV Mono-infection: Exploring Non-invasive Methods for Diagnosis and the Therapeutic Role of Vitamin E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Giada Sebastiani, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNPT 024
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: HIV Mono Infection
MeSH Terms: interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin E intervention (Experimental): All study participants receive Vitamin E 800 IU once daily for 6 months
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin E — Vitamin E 800 IU once daily

SUMMARY:
Effective combination antiretroviral therapy (cART) has resulted in a dramatic reduction in AIDS mortality. Over the last decade, the proportion of deaths caused by liver-related etiologies, including co-infection with hepatitis C (HCV) and hepatitis B (HBV) viruses, alcohol abuse, and fatty liver, has increased between 8 to 10 fold in the post-cART era while AIDS-related mortality has fallen more than 90-fold. HIV infection without viral hepatitis is also at risk for liver disease. Indeed, HIV mono-infected persons experience common conditions, such as obesity, diabetes and dyslipidemia, which are risk factors for non-alcoholic fatty liver disease (NAFLD). NAFLD is the most common liver disease in Canada. It is a fatty infiltration of the liver that is not evolutive per se, but it is the first histopathological step for non-alcoholic steatohepatitis (NASH), a progressive disease characterized by much inflammation leading to liver fibrosis and cirrhosis. NASH may be frequent in the setting of HIV mono-infection due to excess of metabolic risk factors, long-term cART, HIV itself and lipodystrophy. An early diagnosis of NASH is essential to establish a prognosis and initiate interventions to reduce progression of liver disease towards cirrhosis. Early diagnosis of NASH is critical for targeting metabolic and hepatologic interventions, which can impact on progression to cirrhosis and end-stage complications. Non-invasive tools for liver fibrosis and NASH, including Fibroscan/CAP and CK-18, are accurate and ideal for screening and serial monitoring. No study has specifically targeted the non-invasive diagnosis of NASH in HIV mono-infected patients. There has been no study about the use of CK-18 as a biomarker for NASH in the setting of HIV mono-infection. Furthermore, CAP has never been applied to this specific population. Finally, there is no data about the potential beneficial therapeutic effect of vitamin E on NASH associated to HIV infection. The investigators hypothesize that CK-18 and Fibroscan/CAP can be used as non-invasive tests to diagnose NASH in HIV mono-infected persons. Likewise, the investigators hypothesize that there will be a significant prevalence of NASH diagnosed by non-invasive tools among patients with HIV mono-infection. The investigators further hypothesize that a 6 months treatment trial with vitamin E supplementation will improve non-invasive diagnostic tests, and/or the metabolic and hepatic profile in HIV mono-infected patients with a non-invasive diagnosis of NASH.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed positive serology for HIV mono-infection and 18 years or older; valid Fibroscan/CAP;
* Able to provide informed consent, signing forms available in French or English.
* Fatty liver (CAP>237.8 dB/m) AND CK-18 levels > 246 U/L OR
* Fatty liver (CAP>237.8 dB/m) AND CK-18 149 U/L + chronically elevated liver function tests (transaminases) + at least 1 metabolic risk factor (among diabetes, insulin resistance, dyslipidemia or overweight).

Exclusion Criteria:

* Co-infection with HCV or HBV (presence of serum HCV-Ab or HbsAg); HCC, liver transplantation
* Significant alcohol consumption, as per AASLD guidelines on NAFLD: "ongoing or recent alcohol consumption > 21 drinks on average per week in men and > 14 drinks on average per week in women"
* Patients taking anticoagulants (warfarin, heparin)
* Patients undergoing chemotherapy or radiotherapy for cancer
* History of diagnosis of prostate cancer
* Planning to become, suspected to be, pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Improvement of NASH diagnosed by non-invasive methods | 6 months
  Assessed by i) difference in AST and/or ALT
Improvement of NASH diagnosed by non-invasive methods | 6 months
  Assessed by ii) difference in Fibroscan/CAP measurements
Improvement of NASH diagnosed by non-invasive methods | 6 months
  Assessed by iii) difference in CK-18 levels

SECONDARY OUTCOMES:
Change in metabolic markers | 6 months
  HOMA
Change in metabolic markers | 6 months
  Cholesterol or triglyceride levels
Change in metabolic markers | 6 months
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Giada Sebastiani, Principal Investigator — Chronic Viral Illness Service, MUHC
Locations (1):
- Chronic Viral Illness Center at Royal Victoria Hospital in McGill university Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No